CLINICAL TRIAL: NCT03873870
Title: The Clinical Impact of 68Ga-DOTATATE PET in the Management of Patients With Neuroendocrine Tumors
Brief Title: 68Ga-DOTATATE PET for Management of Neuroendocrine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-5034; PET NET Registry (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Neuroendocrine Tumors
Keywords: PET scans
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga -DOTATATE PET scan (Experimental): Single arm study.
  Interventions: Diagnostic Test: 68Ga -DOTATATE PET scans

INTERVENTIONS:
Diagnostic Test: 68Ga -DOTATATE PET scans — PET scan using 68Ga-DOTATATE contrast

SUMMARY:
This is a research study to collect information regarding usefulness of positron emission tomography (PET) scans using a special dye called 68Ga-DOTATATE for patients with neuroendocrine tumours by determining the number of of patients whose clinical management was changed as a result of the scans.

DETAILED DESCRIPTION:
When patients are suspected of having neuroendocrine tumours, they will usually undergo various imaging scans such as computed tomography (CT) scan and magnetic resonance imaging (MRI), and octreotide scintigraphy (octreoscan) to try to identify the primary tumour. During the patients' course of disease, they will continue to have various CT, MRI, and/or octreoscans. Sometimes, despite using scans, laboratory tests, and examination, it is still difficult to properly diagnose neuroendocrine tumours.

Doctors have found that most neuroendocrine tumours make too much of a hormone called somatostatin on their cell surface. Because of this doctors have been using positron emission tomography (PET) scans using a special contrast dye called 68Ga-DOTATATE in hopes of better diagnosing and managing neuroendocrine tumours. 68Ga-DOTATATE can label the cells that have somatostatin (such as neuroendocrine tumour cells) so that the PET scan can take better pictures and doctors can better diagnose and manage the disease.

However, despite 68Ga-DOTATATE PET scans showing promise, it is still not widely accessible. Because of this, researchers are creating a registry for patients who may need 68Ga-DOTATATE PET scans to:

* Identify their primary tumour where the doctor suspects is a neuroendocrine tumour
* Staging of the neuroendocrine tumour
* Restage the tumour prior to surgery/radiotherapy or help to assess the tumour where standard scans such as CTs, MRIs, or octreoscans are not properly showing your tumours despite other clinical or laboratory tests showing that your disease has progressed
* For other issues when confirmation of site of disease and/or disease extent may impact clinical management of the neuroendocrine tumour.

This registry help the participant's treating physician to obtain approval for the participant to undergo 68Ga-DOTATATE PET scans for their neuroendocrine tumour.

ELIGIBILITY:
Inclusion Criteria:

* Able to undergo PET/CT without sedation
* Any of the following indications:

  * Group A. Identification of primary tumor: For the initial diagnosis of patients with clinical (e.g., signs, symptoms) and/or biochemical (e.g., tumor markers) suspicion of neuroendocrine tumours (NETs) but for whom conventional imaging is negative or equivocal or for whom biopsy is not easily obtained.
  * Group B. Staging: For the staging of patients with localized primary NETs and/or limited metastasis where definitive surgery is planned.
  * Group C. Restaging: Restaging of patients with NET where surgery or peptide-receptor radiotherapy (PRRT) is being considered; OR, where conventional imaging is negative or equivocal at time of clinical and/or biochemical progression.
  * Group D. As a problem-solving tool: As a problem-solving tool in patient with NET when confirmation of site of disease and/or disease extent may impact clinical management.
* Approved by a review panel if Group D.

Exclusion Criteria:

* Inability to provide informed consent.
* Contraindication for PET examination as per institutional safety guidelines, including but not limited to pregnancy, or inability to lie still for PET examination.
* Need for full sedation to undergo PET/CT scan.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1916 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Detection of additional disease and/or change in extent of disease after 68Ga-DOTATATE PET | NA. One time visit for 68Ga-DOTATATE PET scan
  Detection of additional disease and/or change in extent of disease after 68Ga-DOTATATE PET

SECONDARY OUTCOMES:
To determine the proportion of patients with NET (or clinical suspicion of NET) in whom intended clinical management prior to PET is changed after 68Ga-DOTATATE PET. | NA. One time visit for 68Ga-DOTATATE PET scan
  To determine the proportion of patients with NET (or clinical suspicion of NET) in whom intended clinical management prior to PET is changed after 68Ga-DOTATATE PET.

CONTACTS AND LOCATIONS:
Overall Officials: Ur Metser, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada